CLINICAL TRIAL: NCT06449157
Title: Chocolate or Sevoflurane: Use of Parosmia to Facilitate More Cooperative Inhalation Inductions in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00434506
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia; Pediatrics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalation induction with parosmia (Experimental): The experimental group will be told about a magical machine that can change the smell of the mask to any flavor the patient desires. The participant will be asked to take a deep breath thinking about that smell and then sevoflurane will be introduced. The patient will be asked if the the chosen flavor is smelled and the response will be noted.
  Interventions: Other: Inhalation induction with parosmia
- Standard inhalation induction (No Intervention): Standard inhalation induction.

INTERVENTIONS:
Other: Inhalation induction with parosmia — The experimental group will then be told that the patient's favorite smell will be put into the face mask via the "magical machine". The patient will be asked to take a deep breath thinking about that smell and then introduce sevoflurane. The patient will be asked if the chosen flavor is smelled and their response will be noted.
  Arms: Inhalation induction with parosmia

SUMMARY:
Children undergoing surgery and anesthesia are often negatively impacted by anxiety and fear in the preoperative period. Routine inhalational anesthetic induction is a unique aspect of pediatric anesthesia. Inhalation inductions are usually initiated with sevoflurane with or without nitrous oxide. While less pungent than other volatile agents, sevoflurane at high concentrations and flows used for inhalation inductions still causes children to often repel from the smell. This can lead to an unpleasant interaction and cause heightened anxiety for any subsequent procedures.

Olfactory senses are processed in the hippocampus and amygdala and tied to emotion and memory. Parosmia is the distortion of smell perception which can utilized to the pediatric anesthesiologists advantage. It has been demonstrated that using this phenomenon, the anesthesiologist can induce a better smell for the child leading to improved cooperation during an inhalation induction. However, limitations of this study include lack of randomization, small sample size, and use of a nominal scale of yes or no for face mask acceptance. The investigators identified no other studies to validate this potentially powerful tool to optimize anesthetic induction for pediatric patients.

The overall objective of this pilot randomized trial is to determine the feasibility of parosmia during inhalation inductions to decrease perioperative stress for children and provide key pilot data to power a larger study to determine effectiveness of parosmia during inhalation inductions to decrease perioperative stress for children and provide key pilot data to power a larger study to determine effectiveness of parosmia.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 5-12 years old
* American Society of Anesthesiologist physical status classification system (ASA) I and II
* Patients coming from home

Exclusion Criteria:

* Patients undergoing emergent surgery
* Patients who have not adequately maintained preoperative nothing per mouth/os (NPO) status
* Patients with inability to communicate verbally
* Tracheostomy patients
* ASA III , IV, V patients

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Perioperative anxiety as assessed by the Modified Yale Preoperative Anxiety Scale-Short Form (mYPAS-SF) | perioperatively
  The modified Yale Preoperative Anxiety Scale-Short Form (mYPAS-SF) will be used to evaluate perioperative anxiety. Patients are evaluated in 4 domains: activity (score 1,2,3, or 4), vocalizations (score 1,2,3,4,5 or 6), emotional expressivity (1,2,3 or 4), and state of apparent arousal (1,2,3, or 4), with higher numbers indicating the highest severity within that item. Each score is calculated by dividing each item rating by the highest possible rating (i.e., 6 for the "vocalizations" item and 4 for all other items), adding all the produced values, dividing by 5, and multiplying by 100. This calculation produces a score ranging from 23.33 to 100, with higher values indicating higher anxiety.

SECONDARY OUTCOMES:
Number of antiemetic mediations administered post-operatively | immediately after the surgery
  Measuring statistical difference in 1) number of antiemetic medications administered
Type and total dose of opioids administered post-operatively | immediately after the surgery
  Type and total dose of opioids administered
Length of time (minutes) to post-anesthesia care unit (PACU) discharge | admission to the PACU through discharge from the PACU (<2 hours post-operatively)
  Length of time from admission to PACU discharge between the control group and the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Pooja O'Neil, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No